CLINICAL TRIAL: NCT00699829
Title: Comparative Medico-Economic Evaluation of Micrographic Mohs Surgery (MMS) and Traditional Surgical Excision With Immediate or Differed Reconstruction to Treat High Recurrence Risk Basal-Cell Carcinomas (BCC)
Brief Title: Mohs Versus Traditional Surgery - Basal-Cell Carcinomas (BCC)
Acronym: BACHIMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Département de la Recherche Clinique, AP-HP
Other Study IDs: P070158
Record Dates: First submitted 2008-05-06; First posted 2008-06-18 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Carcinoma, Basal Cell
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Mohs' micrographic surgery (MMS)
- 2: Conventional surgery

SUMMARY:
Mohs' micrographic surgery (MMS) is a treatment of choice for high recurrence risk basal-cell carcinomas (BCC). Realized under local anaesthesia, it induces very low recurrence rates and spares unnecessary excision of intact surrounding tissues, thus decreasing the needs for flaps, skin grafts, and allows immediate reconstruction…. Its disadvantages are mainly: need for a significant training of the operator, the pathologist and the non-medical personnel; longer duration of the procedure, with higher a priori costs, and constraints for the patient related to the duration of the intervention. Traditional surgical excision with immediate or differed reconstruction is the technique of reference. Provided that re-excisions are performed as long as previous ones do not guarantee free margins, it gives good results. Its real costs are poorly known and can be enhanced by several considerations: multiplicity of the operational acts if the initial excision is insufficient, more complex reconstruction procedures, duration of post-operative dressings, ….

The investigators' objective is to know the costs of the surgical treatment of the high risk CBC, comparing the CMM with the surgical excision with immediate or differed reconstruction, along with its effectiveness defined by the absence of recurrence. by its impact on the quality of life of the patient. It is a prospective, multicentric, comparative, not randomized, open, cohort study, of the type "here and elsewhere". Patients with high-risk CBC, as defined by the French ANAES Guidelines (2004), will be included:

* clinically morpheaform aspect or ill-limited margins, aggressive histological forms;
* already recurred BCC (except for superficial BCCs));
* nodular BCC located in the high-risk zone (nose, peri-orificial areas of the head) and with diameter larger than 1 cm.

The effectiveness will be measured by the rate of recurrence at 5 years (as measured by the prolongation of the follow-up after the surgical procedure). The utility from the patient point of view will be evaluated by a specific dermatologic quality of life questionnaire (Skindex) and by a generic questionnaire (Euroqol 5D), supplemented by a questionnaire of satisfaction of the care (Attkisson). The economic perspectives studied will be those of the hospital, of the payer and of the society. Direct medical costs will be evaluated by micro-costing. The main production factors implied in the realization of one CMM or one traditional surgery in dermatology/surgery and anatomopathology wards will be identified, counted, and developed. The measuring units will be the estimate of the time devoted to each individual procedure, reported to the total activity of each ward and the wages of the various categories of personnel implied, and the unit costs in consumable and redeemable material, reported to their utilisation factor. The hospital indirect costs will be estimated by the financial services of the hospitals. Accrual of 150 CMM and 300 traditional excisions will be performed within a two year period of time.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Histologically proved cutaneous BCC
* Categorized as "bad prognostic" according to the 2004 recommendations of ANAES

  1. morpheaform or ill-limited clinical forms and histologically aggressive forms (morpheaform, micronodular, infiltrating, squamous differentiation) OR
  2. already recurred BCC (except for superficial BCCs) OR
  3. nodular BCCs from the high-risk zone (nose and peri-orificial areas of the head) and with diameter larger than 1 cm.
* Life expectancy greater than 3 years according to the investigator's opinion.
* Patient being informed and having signed the consent to participate to the study

Exclusion Criteria:

* History of X-ray therapy in the territory of the BCC
* Counter-indication to surgery
* Life expectancy < 3 years
* superficial BCCs, even if recurred
* Patient being unable to attend future follow-up visits
* Patient with severe cognitive impairment
* Patient not affiliated to a social security regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients de services de dermatologie et/ou chir plastique
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2008-06

PRIMARY OUTCOMES:
Cost-utility ratio | 2 years

SECONDARY OUTCOMES:
2 and 5 years survival | 2 & 5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Philippe SAIAG, Principal Investigator — Hospital Ambroise Paré Paris; Jean-Marie SERVANT, Principal Investigator — Hôpital Saint Louis
Locations (1):
- Hôpital Ambroise Paré, Boulogne, France